CLINICAL TRIAL: NCT05355974
Title: Vasopressor Utilization to Support Mean Arterial Pressure During Rapid Sequence Intubation: A Clinical Trial (Rapid-Press Trial)
Brief Title: Using Vasopressor Medication to Support Blood Pressure During Intubation Procedure
Acronym: RAPID PRESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2022-43; IRB-2022-43 (Other: Wright State University IRB)
Record Dates: First submitted 2022-04-25; First posted 2022-05-02 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Failure; Hypotension and Shock; Hypotension on Induction; Intubation Complication; Anesthesia Intubation Complication
Keywords: mean arterial pressure; Rapid Sequence Intubation; vasopressor; Norepinephrine; Hypotension from Intubation
MeSH Terms: conditions — Respiratory Insufficiency; Hypotension; Shock | interventions — Norepinephrine; Ringer's Lactate; Saline Solution; Plasma-lyte 148; Plasmalyte A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Norepinephrine plus Isotonic Fluids (Experimental): The treatment group will receive a continuous infusion of norepinephrine at 0.10 mcg/kg/min started 2-5 minutes prior to Rapid Sequence Intubation (assuming normal systolic blood pressure 90-140mmHg) in addition to a standard fluid bolus of Lactated Ringers or Normal Saline or Plasmalyte at 999 mL/hr.
  Interventions: Drug: Norepinephrine; Drug: Lactated Ringers, Intravenous; Drug: normal saline; Drug: Plasma-lyte
- Isotonic Fluids (Active Comparator): The control group will receive an infusion of Lactated Ringers or Normal Saline or Plasma-Lyte with at least 500 mL at 999 ml/hr 2-5 minutes prior to Rapid Sequence Intubation.
  Interventions: Drug: Lactated Ringers, Intravenous; Drug: normal saline; Drug: Plasma-lyte

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine continuous infusion at 0.10 mcg/kg/min
  Other Names: Levophed; Norepinephrine Bitartrate; Norepinephrine-Dextrose
  Arms: Norepinephrine plus Isotonic Fluids
Drug: Lactated Ringers, Intravenous — 500mL infusion run at 999mL/hr
  Other Names: Ringer's Injection; Hartmann's Solution; LR
Drug: normal saline — 500mL infusion run at 999mL/hr
  Other Names: NS; 0.9 percent Sodium Chloride
Drug: Plasma-lyte — 500mL infusion run at 999mL/hr
  Other Names: Plasma-Lyte 148; Plasmalyte

SUMMARY:
The purpose of this study is to investigate whether protocolized vasopressor use for patients with normal blood pressure undergoing rapid sequence intubation improves hemodynamic parameters and mitigates adverse events.

The hypothesis is that use of vasopressors during Rapid Sequence Intubation will prevent substantial decreases in blood pressure when compared to normal intravenous fluids.

DETAILED DESCRIPTION:
Aim: Prevent 25-46 percent reduction in systolic blood pressure associated with rapid sequence intubation with norepinephrine compared to isotonic fluids alone.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory Failure Requiring Intubation

Exclusion Criteria:

* Pregnancy
* Patients intubated during code blue clinical scenarios
* Requiring surgical airway
* Failed intubations
* MAP less than 65 or Systolic Blood Pressure (SBP) less than 90mmHg pre-intubation
* Systolic blood pressure greater than 150mmHg
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 1 hour after Rapid Sequence Intubation
  Change in systolic blood pressure during rapid sequence intubation in mmHg.

SECONDARY OUTCOMES:
Change in serum creatinine (Acute Kidney Injury) | 24 hours after Rapid Sequence Intubation
  Change in serum creatinine (in mL) after rapid sequence intubation and development of Acute Kidney Injury as defined by ≥0.3 mg/dL (≥26.5 micromol/L) within 48 hours
Acute Kidney Injury | 24 hours after Rapid Sequence Intubation
  Change in urine output (in mL) after rapid sequence intubation and development of Acute Kidney Injury as defined by Urine volume <0.5 mL/kg/hour for six hours

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Koroscil, MD, Principal Investigator — Wright State University; Yonatan Dollin, DO, Principal Investigator — Wright State University
Locations (1):
- Miami Valley Hospital Premier Health, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD